CLINICAL TRIAL: NCT06920030
Title: Pilot Study to Investigate the Performance of the Cardiac Microcurrent (C-MIC) System With a Less Invasively Placed Left Ventricular Lead
Brief Title: Performance of the Cardiac Microcurrent (C-MIC) System With a Less Invasively Placed Left Ventricular Lead
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berlin Heals GmbH (Industry)
Collaborators: SCIRENT Clinical Research and Science d.o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C-MIC-III
Record Dates: First submitted 2025-04-01; First posted 2025-04-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Cardiomyopathy; Left Ventricular (LV) Systolic Dysfunction
Keywords: dilated cardiomyopathy; heart failure
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Intervention Model Description: The CMIC-device effect was investigated in previous clinical studies. However, placement of the Left Ventricular Patch Lead up to now requires invasive surgery. This study shall investigate three different procedures with less invasive placement of the LV patch lead.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sub-Q implantation (Experimental): The LV patch electrode will be positioned in a left-thoracic subcutaneous pocket
  Interventions: Device: Subcutaneous cardiac microcurrent treatment
- device-pocket (Experimental): The LV patch electrode will be placed in the same pocket as the device itself
  Interventions: Device: Infraclavicular pocket cardiac microcurrent treatment
- Coronary Sinus placement (Experimental): A coronary sinus electrode will be placed instead of a patch
  Interventions: Device: Coronary Sinus cardiac microcurrent treatment

INTERVENTIONS:
Device: Subcutaneous cardiac microcurrent treatment — An implantable device that emits a weak direct (DC)-microcurrent directly to the heart, using a coil electrode that is transvenously placed in the right ventricle and a patch electrode that is placed in a left thoracic subcutaneous pocket
  Arms: Sub-Q implantation
Device: Infraclavicular pocket cardiac microcurrent treatment — An implantable device that emits a weak direct (DC)-microcurrent directly to the heart, using a coil electrode that is transvenously placed in the right ventricle and a patch electrode that is placed in the same infraclavicular pocket as the device itself
  Arms: device-pocket
Device: Coronary Sinus cardiac microcurrent treatment — An implantable device that emits a weak direct (DC)-microcurrent directly to the heart, using a coil electrode that is transvenously placed in the right ventricle and a coronary sinus electrode
  Arms: Coronary Sinus placement

SUMMARY:
Patients with idiopathic dilative cardiomyopathy in heart failure (NYHA III - IVa) despite adequate therapy according to treatment guidelines and who have a baseline left ventricular ejection fraction between ≥25% and ≤35% will receive a C-MIC treatment together with optimal medical management. The device will be implanted in 3 different ways without the need to open the chest. Each patient will be assigned to one implantation technique. At the end of the study after 6 months, the C-MIC System will be turned off. The primary endpoint of the study is the change in left ventricular ejection fraction after 6 months of treatment.

DETAILED DESCRIPTION:
Target patients for the C-MIC System are patients with idiopathic dilative cardiomyopathy who have systolic left ventricular dysfunction (NYHA class III - NYHA class IV) despite adequate therapy of heart failure and a left ventricular ejection fraction ranging from 25% to 35% with a history of heart failure of more than 1 year but less than 5 years.

In previous studies, C-MIC was successfully implanted with one of the electrodes (the LV patch electrode) being placed directly on the heart with the necessity to perform a thoracotomy.

In this study the the LV patch electrode will be placed in 2 different locations outside of the ribcage so that there is no need to perform a thoracotomy and in a 3rd group, a coronary sinus electrode is placed instead. In group 1, the LV patch electrode will be placed in a left-thoracic position into a subcutaneous pocket. In group 2, the LV patch electrode will be placed into one subcutaneous, infraclavicular pocket together with the microcurrent device itself. In group 3, the LV patch electrode will be replaced with a coronary sinus electrode that is placed transvenously.

In all the groups, the effect of the microcurrent therapy will be assessed by comparing LV election fraction changes between baseline and after 6 months of microcurrent treatment (primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic dilated cardiomyopathy who have systolic left ventricular dysfunction despite adequate therapy of heart failure (NYHA III - IV (ambulatory)).
* Patients with symptomatic chronic heart failure for more than 1 year and less than 5 years at screening based on the date of diagnosis.
* Patients who have a baseline left ventricular ejection fraction of ≥25% and ≤35% assessed by corelab echocardiography within 30 days prior to device implantation.
* Female and male patients aged ≥18 years - 75 years.
* Patient who understands the nature of the procedure and on-going device therapy. Patient is informed about their participation in a chronic clinical trial and about the intended treatment period of 6 months which is derived by the fact that according to current knowledge microcurrent treatment exceeding 6 months will not have additional favorable effects which means it will not further improve cardiac function. Furthermore, the patient is informed about the possibility of device explantation, informed regarding possible risks and is able to give written informed consent prior to any procedures and is considered willing and able to adhere to the study regimen and to return for all followup visits.

Exclusion Criteria:

Patients who are not likely to experience improvement of their chronic heart failure by the microcurrent therapy, because the causes of the disease cannot be influenced even if the patients fulfill the indication for use of the device or if the therapy with the C-MIC System is not possible or might be associated with unknown risks:

* Patients who have a potentially correctible cause of heart failure, such as valvular heart disease or congenital heart disease.
* Patients with an indication for a CRT system according to current guidelines.
* Patients who have been hospitalized for heart failure which required the use of inotropic support within 30 days before screening.
* Patients with systolic blood pressure above 150 mmHg and diastolic blood pressure above 90 mmHg despite optimal antihypertensive medical treatment.
* Patients with hemoglobin blood level < 12 g/dl in male and < 10 g/dl in female patients.
* Patients with primary pulmonary hypertension
* Patients who have genetic connective tissue disease (for example Marfan syndrome).
* Patients with a prosthetic tricuspid valve.
* Patients in whom access for implantation of the leads cannot be obtained (i.e. known venous occlusion, post radiation therapy).
* Patients who have other preexisting epicardial leads.
* Patient with other features (i.e. thorax deformity) that in the eyes of the investigator make the straightforward placement of the device seem unlikely.
* Patients with a pacemaker, an ICD system, a CRT system or with a CCM system*.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception (e.g. intrauterine device, oral contraceptives, barrier methods, or other contraception deemed adequate by the investigator) 2 months before and until 1 month after C-MIC therapy. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 2 months before screening.
* Current pregnancy or
* Breastfeeding/lactating women
* Patients whose exercise tolerance is limited by a condition other than heart failure (e.g. chronic obstructive pulmonary disease, peripheral vascular disease, orthopedic or rheumatologic conditions) or who are unable to participate in a 6-minute walk test.
* Patients on immunosuppressive therapy.
* Patients with present malignancy.
* Patients with an active infection considered by the investigator to be unsafe for the patient's participation in the trial.
* Patients with renal dysfunction (i.e., estimated glomerular filtration rate <45 mL/min /1,73 m²)
* Patients with history or presence of relevant liver diseases or hepatic dysfunction as indicated by abnormal liver function tests at screening and baseline: ALT (SGPT), AST (SGOT), γ-GT, alkaline, phosphatase and serum bilirubin >2 × upper limit of normal (ULN). Increase of these liver enzymes caused by cardiac disorders in the absence of other possible causes of liver damage are not meant by this.
* Patients with a history of drug or alcohol abuse within the 12 months prior to screening.
* Patients who, in the opinion of the Principal Investigator, are unlikely to comply with the protocol requirements, instructions and trial related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits, psychological illness, and improbability of completing the trial.
* Participation in any study of an investigational device or drug within 90 days prior to planned study.
* Vulnerable Patients (e.g. patients requiring a legal representative, patients kept in detention, any service within the army, and employees of the sponsor or at an investigator site).
* Patients who are not able to avoid the following areas (i.e. due to work):

  * Areas with strong magnetic fields
  * Areas with strong external electrical influences
  * Areas with a warning notice "Access prohibited for pacemaker patients" or similar.
  * Areas with high temperatures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
LV ejection fraction change from baseline | 6 months
  Change of LV ejection fraction from baseline to 6 months as measured by echocardiography with Corelab. Difference in means between the two timepoints evaluated separately for each group.

CONTACTS AND LOCATIONS:
Locations (2):
- University Clinical Center of the Republic of Srbska, Banja Luka, Republic of Srbska, Bosnia and Herzegovina
- Institute of Cardiovascular Disease Dedinje, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No